CLINICAL TRIAL: NCT01446991
Title: Phase II Trial Assessing the Feasibility and Toxicity of Degarelix in Achieving Prostate Downsizing Prior to Treatment With Permanent Seed Prostate Brachytherapy
Brief Title: Feasibility and Toxicity of Degarelix for Prostate Downsizing Prior to Permanent Seed Prostate Brachytherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, MD FRCPC Radiation Oncology, British Columbia Cancer Agency
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11-08172
Record Dates: First submitted 2011-10-04; First posted 2011-10-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: prostate neoplasm; brachytherapy; androgen ablation; benign prostatic hypertrophy; prostate size reduction; localized prostate cancer with prostate volume > 40 cc
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Favorable prostate cancer with pubic arch interference (Experimental): Men in this arm have chosen brachytherapy for management of localized prostate cancer and do not require androgen ablation for oncologic reasons but have an enlarged prostate causing pubic arch interference and thus require prostate size reduction prior to brachytherapy. They will have 2-3 months of Degarelix with measurement of prostate volume at 8 and 12 weeks.
  Interventions: Drug: Degarelix
- Intermediate risk prostate cancer, 6 months Degarelix (Experimental): Men in this arm have higher risk prostate cancer (upper tier intermediate risk by National Comprehensive Cancer Network [NCCN] guidelines) and require 6 months of androgen ablation in conjunction with brachytherapy. Prostate size must be > 40 cc at baseline so that prostate size reduction measurements are appropriate. Prostate measurements by transrectal ultrasound with be taken at 12 weeks and 20 weeks.
  Interventions: Drug: Degarelix

INTERVENTIONS:
Drug: Degarelix — 240 mg loading dose followed by monthly 80 mg maintenance dose for 2-3 months
  Arms: Favorable prostate cancer with pubic arch interference
Drug: Degarelix — 240 mg loading dose of Degarelix followed by 80 mg maintenance doses every month for a total duration of 6 months.
  Arms: Intermediate risk prostate cancer, 6 months Degarelix

SUMMARY:
This study will investigate the efficacy of Degarelix, a Luteinizing Hormone Releasing Hormone (LHRH) antagonist, to reduce prostate volume prior to permanent seed prostate brachytherapy. There are 2 eligible populations of men, all of whom will have selected brachytherapy as their treatment of choice for their prostate cancer. Either they have an enlarged prostate that requires size reduction to render brachytherapy technically feasible, or they require androgen ablation in conjunction with brachytherapy for optimal tumor control. The hypothesis is that Degarelix will provide > 30% volume reduction by 3 months in > 30% of men.

DETAILED DESCRIPTION:
All men will have a baseline transrectal ultrasound for brachytherapy planning that has demonstrated an enlarged prostate with or without pubic arch obstruction. After signing the informed consent document they will have a loading dose of 240 mg Degarelix and then monthly maintenance dose injections of 80 mg until such time as sufficient prostate reduction has occured (2-3 months) or they complete the 6 months of required androgen ablation for their disease status.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of prostate cancer
* Favorable risk disease (cT1 or T2a, Gleason score (GS) 6, and Prostate Specific Antigen (PSA) < 10 ng/mL)
* Low-tier intermediate risk disease (cT2c,GS=6,and PSA 10-15 ng/mL, OR GS=7 and PSA < 10 ng/mL)
* Intermediate risk disease AND androgen deprivation therapy recommended by the treating physician for oncologic reasons such as (≥ 50% positive biopsy cores,cT2c,PSA 15-20 ng/mL,GS=7)
* Patient requires baseline planning trans-rectal ultrasound for the purposes of prostate brachytherapy, showing prostate volume > 40 mL and pubic arch interference (not required for those requiring androgen ablation for oncologic reasons)

Exclusion Criteria:

* castrate serum testosterone level
* previous or concurrent pelvic radiotherapy
* unable to give written informed consent
* contraindications to permanent seed prostate brachytherapy or to androgen deprivation therapy
* prior treatment for prostate cancer
* prior trans-urethral resection of the prostate
* previous therapy with a 5-α reductase inhibitor, anti-androgen agent, or LHRH agonist
* previous therapy with degarelix

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-04; Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
prostate volume reduction | 3 months
  determined by transrectal ultrasound with planimetry volume calculation

SECONDARY OUTCOMES:
testosterone recovery | 12 months
  Luteinizing Hormone(LH), Follicle Stimulating Hormone (FSH) and testosterone will be measured at 1, 3, 6, 9 and 12 months following cessation of Degarelix.

CONTACTS AND LOCATIONS:
Overall Officials: Juanita M Crook, MD, Principal Investigator — British Columbia Cancer Agency
Locations (3):
- Canada (3):
  - Abbottsford Cancer Center, Abbottsford, British Columbia
  - Fraser Valley Cancer Center, Surrey, British Columbia
  - Vancouver Cancer Center, Vancouver, British Columbia

REFERENCES:
- [Derived] Korzeniowski MA, Crook JM, Bowes D, Gaztanaga M, Ots A, Jazwal J, Rose J, Tetreault-Laflamme A, Pilote L, Halperin R, Kim D, Petrik D, Araujo C, Bachand F. A Phase II trial of 8 weeks of degarelix for prostate volume reduction: Efficacy and hormonal recovery. Brachytherapy. 2018 May-Jun;17(3):530-536. doi: 10.1016/j.brachy.2017.12.005. Epub 2018 Feb 2. PMID 29398594